CLINICAL TRIAL: NCT03714906
Title: Utility of Pre-Operative Stellate Ganglion Blockade for Pain Control in Unilateral Head and Neck Cancer Surgery
Brief Title: Stellate Ganglion Block in Head and Neck Cancer Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual, lack of benefit between intervention and control arms on interim analysis
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1317655
Record Dates: First submitted 2018-10-19; First posted 2018-10-22 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Head and Neck Cancer; Pain, Postoperative
Keywords: head and neck cancer; pain; analgesia
MeSH Terms: conditions — Head and Neck Neoplasms; Pain, Postoperative; Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients randomized to the Treatment arm will be assigned to receive a stellate ganglion block. While in the hospital after surgery, patients will be given a regimen of scheduled acetaminophen 650 milligrams every 6 hours. Planned treatment of post-operative pain will include the option of requesting oxycodone on an as-needed basis every four hours and IV morphine for breakthrough pain.
  Interventions: Procedure: Stellate ganglion block
- Control (No Intervention): Patients assigned to the Control arm will receive no pre-operative intervention. While in the hospital after surgery, these patients will be given a regimen of scheduled acetaminophen 650 milligrams every 6 hours. Planned treatment of post-operative pain will include the option of requesting oxycodone on an as-needed basis every four hours and IV morphine for breakthrough pain.

INTERVENTIONS:
Procedure: Stellate ganglion block — Stellate ganglion block will consist of an injection of 0.25% bupivacaine placed under ultrasound guidance by a trained anesthesiologist in the pre-operative holding area prior to surgery.
  Arms: Treatment

SUMMARY:
The purpose of this study is to evaluate and reduce pain and improve quality of life in patients being treated for head and neck cancer with unilateral surgery. In this study, patients will be randomly assigned to receive either pre-operative stellate ganglion block or no pre-operative treatment. Blocks will be placed by a trained anesthesiologist using ultrasound guidance in the preoperative holding area prior to surgery. All patients will receive the same post-operative pain medication regimen with appropriate pain treatment as needed. Patients will be asked to fill out surveys prior to surgery, while in the hospital after surgery, and at each follow-up appointment for up to 24 months.

DETAILED DESCRIPTION:
Sympathetic blockade of the stellate ganglion is used for upper limb, temporomandibular joint, and facial pain, and may be placed pre-operatively to decrease post-operative pain in upper limb orthopedic surgery. Use of this block for head and neck cancer pain has been studied with mixed results in a case series in the distant past prior to the advent of image guidance or newer long-lasting anesthetic drugs. One recent case report for intractable head and neck cancer pain demonstrated encouraging results with relief provided after diagnostic stellate ganglion blockade followed by chemical neurolysis.

Patients who choose to participate in the study will be randomly assigned to receive either stellate ganglion block placement in the pre-operative holding area on the day of surgery or no pre-operative intervention. Participating patients will be asked to fill out separate questionnaires to evaluate pain and quality of life preoperatively and post-operatively.

Upon enrollment in the study, patients will be assigned an identification number and will undergo simple randomization to either the control or treatment group using a randomly computer-generated sequence. If patients have not had an evaluation of vocal cord mobility on prior workup, this will be assessed by flexible fiberoptic laryngoscopy prior to proceeding with block placement.

Patients assigned to receive a block will have it placed on the respective surgical side in the pre-operative holding area on the day of surgery. A trained anesthesiologist will perform the placement using an injection of 0.25% bupivacaine under ultrasound guidance. While in the hospital after surgery, patients will be given a regimen of scheduled acetaminophen 650 milligrams every 6 hours. Planned treatment of pain will include the option of requesting oxycodone on an as-needed basis every four hours and IV morphine for breakthrough pain. Surveys will be administered and collected on a daily basis while patients are in the hospital. If patients are already utilizing other non-opioid pain medications like muscle relaxers (Flexeril, baclofen, etc.), or neuropathic pain medications (Neurontin), they will be allowed to continue these medications while inpatient provided there are no changes in dosing. Home non-steroidal anti-inflammatory analgesic medications will be withheld while patients are in the hospital due to the potential risk of post-operative bleeding and kidney injury related to use of these medications in the perioperative setting. These medications may be resumed once you are discharged from the hospital.

Patients will be discharged home on a seven-day course of acetaminophen with as-needed oxycodone. Outcomes surveys will then be collected at each subsequent post-operative follow up. Follow up visits will occur one week after discharge, four weeks after discharge, and then every three months until completion of the two year study period.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients who are greater than eighteen years of age with a known diagnosis of head and neck cancer and are planned to undergo surgery with unilateral neck dissection will be eligible for this study

Exclusion Criteria:

* Patients with a history of preoperative narcotic use for conditions unrelated to their head and neck cancer will be excluded.
* Patients younger than eighteen years of age, patients with a history of vocal cord paralysis on the non-surgical side, patients with a history of severe difficulty swallowing, and pregnant patients will be excluded from this study.
* Patients with a history of abnormal heart rhythm will be considered to have a relative contraindication and will require clearance by the consultant anesthesiologist prior to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | 2 years
  Validated pain survey in head and neck cancer patients

SECONDARY OUTCOMES:
Inpatient morphine equivalents | 1-7 days or longer depending on length of stay
  Requirement of short-term post-operative narcotic therapy
Defense & Veterans Pain Rating Scale | 2 years
  Non-validated pain survey in head and neck cancer patients
University of Washington Quality of Life Scale Version 4 (UW-QOL 4) | 2 years
  Validated quality of life outcomes scale in head and neck cancer patients
EuroQol 5D-5L | 2 years
  Non-validated quality of life survey in head and neck cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: James K Byrd, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University Department of Otolaryngology-Head and Neck Surgery, Augusta, Georgia, United States

REFERENCES:
- [Background] Gunduz OH, Kenis-Coskun O. Ganglion blocks as a treatment of pain: current perspectives. J Pain Res. 2017 Dec 14;10:2815-2826. doi: 10.2147/JPR.S134775. eCollection 2017. PMID 29276402
- [Background] Wang QX, Wang XY, Fu NA, Liu JY, Yao SL. Stellate ganglion block inhibits formalin-induced nociceptive responses: mechanism of action. Eur J Anaesthesiol. 2005 Dec;22(12):913-8. doi: 10.1017/S0265021505001559. PMID 16318661
- [Background] McDonnell JG, Finnerty O, Laffey JG. Stellate ganglion blockade for analgesia following upper limb surgery. Anaesthesia. 2011 Jul;66(7):611-4. doi: 10.1111/j.1365-2044.2011.06626.x. Epub 2011 May 31. PMID 21627622
- [Background] Jones GP, Tripathi SS. Successful use of stellate ganglion block and a new centrally acting analgesic with dual mode of action in a resistant temporomandibular joint pain. BMJ Case Rep. 2014 May 20;2014:bcr2013203308. doi: 10.1136/bcr-2013-203308. PMID 24849638
- [Background] Salvaggio I, Adducci E, Dell'Aquila L, Rinaldi S, Marini M, Zappia L, Mascaro A. Facial pain: a possible therapy with stellate ganglion block. Pain Med. 2008 Oct;9(7):958-62. doi: 10.1111/j.1526-4637.2008.00515.x. PMID 18950449
- [Background] Kumar N, Thapa D, Gombar S, Ahuja V, Gupta R. Analgesic efficacy of pre-operative stellate ganglion block on postoperative pain relief: a randomised controlled trial. Anaesthesia. 2014 Sep;69(9):954-660. doi: 10.1111/anae.12774. Epub 2014 Jul 7. PMID 25040168
- [Background] Ghai A, Kaushik T, Kumar R, Wadhera S. Chemical ablation of stellate ganglion for head and neck cancer pain. Acta Anaesthesiol Belg. 2016;67(1):6-8. PMID 27363209